CLINICAL TRIAL: NCT02202096
Title: A Pilot Randomized Trial of the Comprehensive Transitional Care Program for Medically Underserved Colorectal Cancer Surgery Patients
Brief Title: A Pilot Randomized Trial of a Comprehensive Transitional Care Program for Colorectal Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources were not readily available to begin the study.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lillian Kao, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel
Other Study IDs: HSC-MS-13-0336
Record Dates: First submitted 2014-05-19; First posted 2014-07-28 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer; Comprehensive Transitional Care Program
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (plus usual care) (Experimental): Patient education: One-on-one visit Discharge planning: Assessment of barriers to discharge Medication reconciliation: Patient medication review Appointment before discharge: Additional measure to ensure awareness of next clinic visit Transition coach Patient-centered discharge instructions: Enhanced Provider continuity: Specific surgeons responsible for coordinating care with medical/radiation oncology Timely follow-up: Barriers to clinic follow-up visits will be discussed Timely PCP communication Follow-up telephone call Patient hotline: 24 hour follow-up following call to Ask My Nurse number
  Interventions: Other: Patient education: One-on-one visit; Other: Discharge planning: Assessment of barriers to discharge; Other: Medication reconciliation: Patient medication review; Other: Appointment before discharge: Additional measure to ensure awareness of next clinic visit; Other: Transition coach; Other: Patient-centered discharge instructions: Enhanced; Other: Provider continuity: Specific surgeons responsible for coordinating care with medical/radiation oncology; Other: Timely follow-up: Barriers to clinic follow-up visits will be discussed; Other: Timely PCP communication; Other: Follow-up telephone call; Other: Patient hotline: 24 hour follow-up following call to Ask My Nurse number
- Usual Care (No Intervention): Usual care-Standard of care that all colorectal cancer patients normally receive

INTERVENTIONS:
Other: Patient education: One-on-one visit — The navigator or surgeon will have a one-on-one visit with he patient to answer any questions.
  Arms: Intervention (plus usual care)
Other: Discharge planning: Assessment of barriers to discharge — Case management will be consulted on the day of surgery. The navigator will perform an assessment of barriers to discharge based on one-on-one interviews with the patient.
  Arms: Intervention (plus usual care)
Other: Medication reconciliation: Patient medication review — The navigator will review the patient's medications with him/her prior to discharge.
  Arms: Intervention (plus usual care)
Other: Appointment before discharge: Additional measure to ensure awareness of next clinic visit — Additional measures to ensure that patients are aware of the date, time, and place of their clinic visit(s) may include a phone calls or text messages to patients and their caregivers by the navigator, surgeon or clinic nurse.
  Arms: Intervention (plus usual care)
Other: Transition coach — The navigator will assist with coordination of care and tracking follow-up appointments and tests.
  Arms: Intervention (plus usual care)
Other: Patient-centered discharge instructions: Enhanced — Enhanced, language-specific, discharge instructions will be developed and provided to all patients verbally and in a written format designed for patients with limited literacy skills.
  Arms: Intervention (plus usual care)
Other: Provider continuity: Specific surgeons responsible for coordinating care with medical/radiation oncology — Drs. Stefanos Millas (colorectal surgery) and Curtis Wray (surgical oncology) will be responsible for coordinating care with medical and radiation oncology as well as consulting when patients are readmitted to the hospital (if not admitted to the surgical service). Changes will be made to the clinic scheduling process for colorectal cancer surgery patients to minimize wait times, to allow them to be seen on a "walk-in" basis, and to prioritize visits for patients with urgent problems as identified by follow-up calls or inquiries to the Ask My Nurse hotline.
  Arms: Intervention (plus usual care)
Other: Timely follow-up: Barriers to clinic follow-up visits will be discussed — Patients will be queried about financial barriers to clinic follow-up such as lack of money for parking and/or lack of transportation; parking vouchers and taxi/bus vouchers may be provided.
  Arms: Intervention (plus usual care)
Other: Timely PCP communication — The operating surgeon will phone the PCP prior to and upon discharge to discuss concerns and follow-up care plans. Communication via the electronic medical record (EPIC) will also be sent. If the patient does not have a PCP, a referral will be made prior at the initial clinic visit and one provided.
  Arms: Intervention (plus usual care)
Other: Follow-up telephone call — Patients will be contacted by phone by the navigator or surgeon on post-discharge day 1 to identify and address any concerns. If there are concerns, calls may be made on subsequent post-operative days.
  Arms: Intervention (plus usual care)
Other: Patient hotline: 24 hour follow-up following call to Ask My Nurse number — Follow-up will occur within 24 hours of calling the Ask My Nurse number. Patients with emergent problems will be seen immediately by the surgical oncology team if available or the on call surgery team. Patients with non-urgent matters will be called by a member of the surgical oncology team. Arrangements will be made to see the patient in clinic or the ER within the next 8-16 hours depending upon severity and time of day.
  Arms: Intervention (plus usual care)

SUMMARY:
The primary hypothesis is that a comprehensive transitional care program based on the premise of a patient-centered medical home versus routine care reduces emergency room visits and hospital readmissions without increasing costs among cancer patients undergoing surgery at a large safety-net hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer
* Adults, Age 18 years or older
* Undergoing surgery for either palliative cure or palliation

Exclusion Criteria:

* Patients not expected to survive hospital based on the operating surgeon's opinion
* Children under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of post-operative ER visits and readmissions | up to 30 days postoperatively
  The number of times the patient returned to the ER and/or was readmitted to the hospital withing 30 days following their surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States